CLINICAL TRIAL: NCT02892994
Title: Immediate Effect of Ultrasound Therapy on Bilateral Masseter Myalgia: A Randomized Double Blinded Investigational Trial
Brief Title: Immediate Effect of Ultrasound Therapy on Bilateral Masseter Myalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, W.D.McCall, Jr., Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ultrasound Project #2
Record Dates: First submitted 2016-05-06; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: therapeutic ultrasound
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Subjects will receive 5 minutes of ultrasound treatment at 0.4 W/cm^2 and 100% duty cycle on each masseter muscle.
  Interventions: Other: ultrasound
- Placebo (Placebo Comparator): Subjects will receive 5 minutes of ultrasound treatment at zero power on each masseter muscle.
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound

SUMMARY:
This study will compare ultrasound 0.4 W/cm^2 and 100% duty cycle versus no ultrasound (placebo) for bilateral masseter myalgia in up to 38 adult women. The dose will be applied for 5 minutes on each side. Both the dose and the starting side will be randomized. Both the subject and ultrasound operator will be blind to the dose. The outcome measures will be pressure pain threshold on both masseter muscles and both temporalis muscles, self reported pain scale (0, no pain to 10, worst pain ever), thermographic temperature of the muscles, and intraoral temperature. These outcome measures will be taken before and after each dose, so three times per subject.

ELIGIBILITY:
Inclusion Criteria:

Adult females Bilateral myalgia based on Diagnostic Criteria for TMD (DC-TMD) (Schiffman, et al., 2014) Current pain intensity ≥4 out of 10, (where 0 is no pain and 10 is the worst pain ever) on both sides.

Exclusion Criteria:

History or diagnosis of systemic musculoskeletal disorders. Rheumatologic diseases (e.g. fibromyalgia, muscular atrophy). Certain conditions such as neoplasms or fractures. Neuropathies or neurological disorders. Currently taking muscle relaxants or analgesics. Any form of physical therapy within the last 60 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold, change from pre- to post-ultrasound dose. | Immediate. Data taken before and after each dose, so three times in the one session which lasts about one hour to completion..
  The change in pressure pain threshold from before to after the ultrasound (or placebo) will be averaged over the two masseter muscles, and over the two temporalis muscles.
Self reported pain scale, change from pre- to post-ultrasound dose which lasts about one hour to completion. | Immediate. Data taken before and after each dose, so three times in the one session.
  The change in self reported pain scale from before to after the ultrasound (or placebo) will be averaged over the two masseter muscles, and over the two temporalis muscles.
Intraoral temperature | Immediate. Data taken before and after each dose, so three times in the one session which lasts about one hour to completion.
  The intraoral temperature in the buccal area near the masseter muscle will be recorded before and after the ultrasound
Thermographic temperature of the muscles | Immediate. Data taken before and after each dose, so three times in the one session which lasts about one hour to completion.
  The thermographic temperature of each masseter and each temporalis muscle will be recorded before and after the ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Willard McCall, Ph. D., Principal Investigator — SUNY Buffalo
Locations (1):
- School of Dental Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784